CLINICAL TRIAL: NCT04620655
Title: RD13-01 for Patients With r/r CD7+ T-ALL/T-LBL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Min Xiang (Other)
Responsible Party: Sponsor-Investigator, Min Xiang, Professor, Hebei Yanda Ludaopei Hospital
Organization: Hebei Yanda Ludaopei Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHCT-RD13-01-03
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: T Acute Lymphoblastic Leukemia; T-lymphoblastic Lymphoma
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RD13-01 cell infusion (Experimental)
  Interventions: Drug: RD13-01 cell infusion

INTERVENTIONS:
Drug: RD13-01 cell infusion — Universal CAR-T cells targeting CD7

SUMMARY:
This study is designed to explore the safety of RD13-01 for patients with CD7+ relapsed and/or refractory T cell acute lymphoblastic leukemia or lymphoblastic lymphoma. And to evaluate the efficacy and pharmacokinetics of RD13-01 in patients.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 3 to 70 years.
2. Diagnosis of r/r T-ALL/T-LBL.
3. ECOG: 0-2.
4. Life expectancy greater than 12 weeks.
5. Cardiac left ventricle ejection fraction ≥50%.
6. Informed consent explained to, understood by and signed by the patient/ guardian. Patient/guardian is given a copy of informed consent.

Exclusion Criteria:

1. Pregnant or lactating.
2. Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive and peripheral blood hepatitis B virus (HBV) DNA titer detection is not within the normal range; hepatitis C virus (HCV) antibody positive and peripheral blood hepatitis C Viral (HCV) RNA positive; human immunodeficiency virus (HIV) antibody positive; cytomegalovirus (CMV) DNA positive; syphilis positive.
3. Patients with graft-versus-host disease (GVHD) or who need to use immunosuppressive drugs.
4. Participated in other clinical studies within 2 weeks prior to screening.
5. History of alcoholism, drug abuse or mental illness.
6. Any situations that the investigator believes may increase the risk of patients or interfere with the results of study.

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-11-15 (Estimated); Primary Completion 2021-11-15 (Estimated); Study Completion 2022-11-15 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | 4 weeks after infusion

CONTACTS AND LOCATIONS:
Overall Officials: Xian Zhang, Principal Investigator — Hebei Yanda Ludaopei Hospital
Locations (1):
- Hebei Yanda Ludaopei Hospital, Langfang, Hebei, China